CLINICAL TRIAL: NCT07355309
Title: Longer-term Effects of High-dairy Food Patterns on the Gut-brain Axis in Adults With Overweight or Obesity
Brief Title: High-Dairy Food Patterns and Gut-Brain Axis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: National Dairy Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: METC25-043
Record Dates: First submitted 2025-12-10; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Brain Insulin Sensitivity; Brain Vascular Function; Cerebral Blood Flow; Cognitive Performance; Appetite Control; Gut Microbiota

STUDY DESIGN:
Intervention Model Description: This study is a randomized, controlled, crossover intervention trial. Each participant will complete two 8-week intervention periods (high-dairy and low-dairy food patterns) separated by a washout period of at least 8 weeks, resulting in a total study duration of approximately 24 weeks.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): High-Dairy Food Pattern
  Interventions: Dietary Supplement: High-dairy food pattern
- Control (Placebo Comparator): Low-Dairy Food Pattern
  Interventions: Dietary Supplement: Low-dairy food pattern

INTERVENTIONS:
Dietary Supplement: High-dairy food pattern — During the high-dairy period, participants will be instructed to consume 4-5 daily servings of dairy products, including: 1-2 servings of yogurt or cottage cheese (200 mL per serving, ≤1.5% fat), 1-2 servings of milk or buttermilk (250 mL per serving, ≤1.5% fat), and 1-2 servings of cheese (20 g per serving, 20+ or 30+ reduced-fat options).
  Arms: Experimental
Dietary Supplement: Low-dairy food pattern — During the low-dairy control period, participants will restrict dairy intake to a maximum of one serving per day
  Arms: Control

SUMMARY:
Disturbances in brain insulin sensitivity are associated not only with obesity and type 2 diabetes, but also with brain aging and cognitive decline. Longitudinal studies suggest that dietary patterns, particularly those high in dairy intake, may impact brain function via the gut-brain axis. Indeed, dairy foods are known to modulate gut microbiota and may, through this pathway, not only improve brain insulin sensitivity and cognitive performance, but also mental health and appetite regulation. However, underlying mechanisms remain largely unexplored. The primary objective of this study is to evaluate, in older adults with overweight or obesity, the effects of a high-dairy food pattern (4-5 daily servings of (butter)milk, cheese, yogurt, or cottage cheese) compared to a low-dairy food pattern (≤1 serving daily) on (regional) brain vascular function and insulin sensitivity. These outcomes will be quantified using the non-invasive MRI perfusion technique Arterial Spin Labeling (ASL), which assesses cerebral blood flow (CBF) in response to intranasal insulin, a validated physiological marker of brain insulin sensitivity. Secondary objectives include changes in cognitive performance (via the CANTAB neuropsychological test battery), gut microbiota composition (via shotgun metagenomic analysis of fecal samples), and appetite-related brain reward activity (via BOLD-fMRI with food cues). Exploratory analyses include conventional cardiometabolic risk markers (blood pressure, lipid and glucose metabolism), and perceivable (consumer) benefits.

ELIGIBILITY:
Inclusion Criteria:

* Men and postmenopausal women (≥ 2 years since last menstruation);
* Aged between 40-75 years;
* BMI between 25-35 kg/m2 (overweight or obese);
* Low-to-moderate habitual dairy consumption (≤ 3 servings/day);
* Fasting serum total cholesterol < 8.0 mmol/L;
* Fasting serum triacylglycerol < 4.5 mmol/L;
* Fasting plasma glucose < 7.0 mmol/L;
* Systolic blood pressure < 160 mmHg and diastolic blood pressure < 100 mmHg;
* Stable body weight (weight gain or loss < 3 kg in the past three months).

Exclusion Criteria:

* Left-handedness;
* Milk protein allergy or lactose intolerance;
* Current smoker, or smoking cessation < 12 months;
* Familial hypercholesterolemia;
* Abuse of drugs;
* Alcoholic intake >3 standard drinks/day;
* Use of medications, food products or dietary supplements affecting glucose, lipid, or blood pressure regulation, gut microbiota or mental or neurological function, judged by the principal investigator;
* Use of antibiotics within the previous month;
* Use of other biomedical investigational products within the previous month;
* Participation in another clinical trial within the past month;
* Severe medical conditions including type 2 diabetes, epilepsy, asthma, kidney failure, COPD, inflammatory bowel disease, autoimmune diseases, or rheumatoid arthritis;
* History of cardiovascular events (e.g., heart attack, stroke) or active cardiovascular disease;
* Contra-indications for MRI imaging (e.g. pacemaker, metal implants, claustrophobia);
* Willing to donate blood starting from 8 weeks before the study begins, throughout the study, and for 4 weeks after its inclusion;
* Difficult to venipuncture as evidenced during the screening visit.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-22 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Brain Insulin Sensitivity | Change in brain insulin sensitivity (difference in CBF [mL/100 g tissue/min] before and after intranasal insulin) at the end of an 8-week high-dairy food pattern and an 8-week low-dairy food pattern
  Cerebral blood flow measurements before and after a nasal insulin spray as quantified non-invasively by the MRI perfusion method Arterial Spin Labeling (ASL)
Brain vascular function | Change in brain vascular function (CBF in mL/100 g tissue/min) at the end of an 8-week high-dairy food pattern and an 8-week low-dairy food pattern
  Cerebral blood flow as quantified non-invasively by the MRI perfusion method Arterial Spin Labeling (ASL)

SECONDARY OUTCOMES:
Cognitive Performance | Change in cognitive performance (test-specific standardized scores) at the end of an 8-week high-dairy food pattern and an 8-week low-dairy food pattern
  Cambridge Neuropsychological Test Automated Battery (CANTAB)
Gut microbial composition | Change in gut microbial composition (shannon index indicating α-diversity) using gene relative abundance profiles at the start and end of an 8-week high-dairy food pattern and an 8-week low-dairy food pattern
  Shotgun metagenomics of fecal samples
Appetite-related brain reward activity | Change in appetite-related brain reward activity (functional connectivity [BOLD signal changes]) at the end of an 8-week high-dairy food pattern and an 8-week low-dairy food pattern
  Appetite-related brain reward activity will be assessed by blood oxygenation level-dependent (BOLD) functional MRI responses to standardized food cues

OTHER OUTCOMES:
Office blood pressure | Change in blood pressure (in mmHg) at the end of an 8-week high-dairy food pattern and an 8-week low-dairy food pattern
  Office blood pressure
Heart rate | Change in heart rate (in beats/min) at the end of an 8-week high-dairy food pattern and an 8-week low-dairy food pattern
  Heart rate
Glucose concentrations | Change in circulating glucose concentrations (in mmol/L) at the end of an 8-week high-dairy food pattern and an 8-week low-dairy food pattern
  Circulating glucose concentrations
Insulin concentrations | Change in insulin concentrations (in mIU/L) at the end of an 8-week high-dairy food pattern and an 8-week low-dairy food pattern
  Circulating insulin concentrations
Lipid metabolism | Change in circulating lipid concentrations (in mmol/L) at the end of an 8-week high-dairy food pattern and an 8-week low-dairy food pattern
  Circulating lipid concentrations
Markers related to low-grade systemic inflammation | Change in circulating high-sensitive C-reactive protein concentrations (in mg/dl) at the end of an 8-week high-dairy food pattern and an 8-week low-dairy food pattern
  Circulating high-sensitive C-reactive protein concentrations
Perceived hunger | Change in perceived hunger (in mm) at the end of an 8-week high-dairy food pattern and an 8-week low-dairy food pattern
  Visual analogue scale (VAS) questionnaires for hunger
Perceived satiety | Change in perceived satiety (in mm) at the end of an 8-week high-dairy food pattern and an 8-week low-dairy food pattern
  Visual analogue scale (VAS) questionnaires for satiety
Perceived desire to eat | Change in perceived desire to eat (in mm) at the end of an 8-week high-dairy food pattern and an 8-week low-dairy food pattern
  Visual analogue scale (VAS) questionnaires for desire to eat
Perceived fullness | Change in perceived fullness (in mm) at the end of an 8-week high-dairy food pattern and an 8-week low-dairy food pattern
  Visual analogue scale (VAS) questionnaires for fullness
Perceived quality of life | Change in perceived quality of life (average score) at the end of an 8-week high-dairy food pattern and an 8-week low-dairy food pattern
  32-item quality of life questionnaire to assess perceived quality of life
Perceived mood | Change in perceived mood (average score) at the end of an 8-week high-dairy food pattern and an 8-week low-dairy food pattern
  Affect Grid Questionnaire to assess perceived mood
Perceived depression and anxiety symptoms | Change in perceived depression and anxiety symptoms (average scores) at the end of an 8-week high-dairy food pattern and an 8-week low-dairy food pattern
  Beck Depression and Anxiety Inventories to assess perceived depression and anxiety symptoms
Perceived stress | Change in perceived stress (average score) at the end of an 8-week high-dairy food pattern and an 8-week low-dairy food pattern
  Perceived Stress Scale questionnaire to assess perceived stress
Perceived sleep quality | Change in perceived sleep quality (average score) at the end of an 8-week high-dairy food pattern and an 8-week low-dairy food pattern
  Pittsburgh Sleep Quality Index to assess perceived sleep quality
Food intake | Change in food intake at the end of an 8-week high-dairy food pattern and an 8-week low-dairy food pattern
  Food Frequency Questionnaire to assess food intake over the past month
Urinary calcium | Change in urinary calcium (mmol/24 hours) at the start and end of an 8-week high-dairy food pattern and an 8-week low-dairy food pattern
  24-hour urine samples for analysis of calcium concentrations
Urinary urea | Change in urinary urea (mmol/24 hours) at the start and end of an 8-week high-dairy food pattern and an 8-week low-dairy food pattern
  24-hour urine samples for analysis of urea concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Ronald P Mensink, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands